CLINICAL TRIAL: NCT04524949
Title: A Phase IIa, Randomized, Double-blind, Dose Comparison, Placebo-controlled, Multi-centre Clinical Trial to Evaluate the Immune Signature of the Treatment With the Imotope IMCY-0098 and Its Effect on the Preservation of Beta-cell Function in Adult Patients With a Recent Onset Type 1 Diabetes
Brief Title: IMCY-0098 Proof of ACtion in Type 1 Diabetes (IMPACT Study)
Acronym: IMPACT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No efficacy at primary analysis after 1 year. Long term follow-up stopped
Sponsor: Imcyse SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMCY-T1D-003; 2020-001317-20 (EudraCT Number)
Record Dates: First submitted 2020-08-11; First posted 2020-08-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus Type 1; Autoimmune disease; Immunotherapy; Diabetes treatment
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- IMCY-0098, low dose (Experimental): The dose A (Cohort 1) will consist of subcutaneous administrations of 450 µg of the peptide in two separate injections of 225 µg each (500 µL each).
  Interventions: Drug: IMCY-0098 450 μg
- IMCY-0098, high dose (Experimental): The dose B (Cohort 2) will consist of subcutaneous administrations of 1350 µg of the peptide in two separate injections of 675 µg each (500 µL each).
  Interventions: Drug: IMCY-0098 1350 μg
- Placebo (Placebo Comparator): Participants randomized to placebo will receive subcutaneous administrations of identical volumes of placebo solution to maintain study blind.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IMCY-0098 450 μg — Small synthetic peptide for SC admin. Solvent: alum hydroxide
  Other Names: Imotope
  Arms: IMCY-0098, low dose
Drug: IMCY-0098 1350 μg — Small synthetic peptide for SC admin. Solvent: alum hydroxide
  Other Names: Imotope
  Arms: IMCY-0098, high dose
Drug: Placebo — Solvent: alum hydroxide
  Arms: Placebo

SUMMARY:
The IMPACT study is a study to test a new experimental drug, IMCY-0098, for the treatment of type 1 diabetes (T1D).

In most people with type 1 diabetes, the pancreas loses its ability to make insulin because some cells of the body's own immune system mistakenly attack and destroy the cells in the pancreas that produce insulin (islet beta-cells).

The study drug IMCY-0098 is being developed to stop the body's own immune system attacking and destroying the insulin-producing cells. When injected, it will induce new immune cells that will specifically destroy the bad immune cells responsible for the damage to the pancreas.

IMCY-0098 has previously been tested on recently diagnosed type 1 diabetes patients in the first clinical study between 2017 and 2019 to collect information on the safety of IMCY-0098. The next step is to test the best dose and the best number of injections that show the drug can give a benefit. Two doses of IMCY-0098 will be tested and they will be compared to a placebo. Safety information will also be collected during the study for all the participants.

DETAILED DESCRIPTION:
The main study will include 84 HLA DR4+ patients. In addition, up to 24 HLA DR4-/DR3+ patients will be included in a mechanistic substudy.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent.
2. Participants aged ≥ 18 years and < 45 years at the time of consent
3. Have a diagnosis of T1D within maximum 9 weeks at screening (date of the first insulin injection)
4. Must have at least one or more diabetes-related autoantibodies present at screening (GAD65, IA-2, or ZnT8)
5. Must have random C-peptide levels ≥ 200 pmol/L measured at screening
6. Must be Human Leukocyte Antigen (HLA) DR4 positive to participate in the main study OR HLA DR4 negative but HLA DR3 positive to participate in the substudy
7. Be willing to comply with intensive diabetes management
8. Be treated with insulin therapy in accordance with the local standard of care
9. Males with reproductive potential must agree to use adequate contraception up to 90 days after the completion of the last treatment. This includes:

   * Barrier contraception (condom and spermicide) or
   * True abstinence (where this is in accordance with the participants preferred and usual lifestyle)
10. All females must have a negative serum pregnancy test at screening. Women sexually active and of childbearing potential must agree to use a highly effective contraception method from screening up to 90 days after last treatment with the investigational product
11. (US ONLY) Have HbA1c levels ≤ 9.5% prior to randomization

Exclusion Criteria:

1. Clinically significant abnormal full blood count (FBC), renal function or liver function at screening including

   1.1. Be immunodeficient or have any clinically significant chronic lymphopenia: Leukopenia (< 3,000 leukocytes /μL), neutropenia (<1,500 neutrophils/μL), lymphopenia (<800 lymphocytes/μL), or thrombocytopenia (<100,000 platelets/μL)

   1.2. Evidence of renal dysfunction with serum creatinine greater than 1.5 times the upper limit of normal OR (US ONLY) estimated Glomerular Filtration Rate (eGFR) calculated by Chronic Kidney Disease Epidemiology Collaboration (CKD-Epi) <90 mL/min per 1.73 m2 in absence of other signs of CKD or rapidly progressing renal disease

   1.3. Evidence of liver dysfunction with aspartate aminotransferase (AST) or alanine transaminase (ALT) greater than 3 times the upper limits of normal or (US ONLY) total bilirubin ≥ 2x Upper Limit of Normal (ULN) or Alkaline phosphatase ≥ 2x ULN. For participants presenting with values above ULN but below above threshold for these parameters, the underlying reason should be investigated by the site team to exclude liver disease. Patients for which a liver disease would be diagnosed will be excluded from the study.

   Participants with elevated unconjugated bilirubin (Gilbert's syndrome) are eligible if bilirubin is ≤ 3 times the upper limits of normal and hepatic enzymes and function are otherwise normal (AST/ALT/Alkaline phosphatase within ULN), and there is no evidence of hemolysis
2. Have signs or symptoms of serious active infection requiring IV antibiotics and/or hospitalization at study entry
3. Have signs or symptoms of active COVID infection or a positive COVID PCR test during the screening period
4. Have received any live attenuated vaccine within 3 months prior to the first planned administration of the study product (which includes, but is not limited to: oral poliomyelitis vaccine, measles-mumps-rubella vaccine, yellow fever vaccine, Japanese encephalitis vaccine, dengue vaccine, rotavirus vaccine, varicella vaccine, live-attenuated zoster vaccine, Bacillus Calmette-Guérin [BCG] vaccine, oral typhoid vaccine)
5. Be currently pregnant or lactating, or anticipate getting pregnant until at least 24 weeks after last study drug administration
6. Require the use of immunosuppressive agents including chronic use of systemic steroids. Topical, inhalational or intranasal corticosteroids are allowed
7. Have evidence of current or past human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C infection
8. Presence of any uncontrolled disease (including uncontrolled autoimmune disease) or abnormal clinical laboratory results that may interfere with study conduct as judged by the investigator
9. History of, or current malignancy (except excised basal cell skin cancer)
10. Current or ongoing use of non-insulin pharmaceuticals that affect glycaemic control within 7 days prior to screening visit
11. Active participation in another T1D treatment study or any investigational intervention study in the previous 30 days or (US ONLY) received gene therapy in the past
12. Known hypersensitivity to any component of the drug product
13. CRO or Sponsor employees or employees under the direct supervision of the Investigator and/or involved directly in the study
14. Be diagnosed with Latent Autoimmune Diabetes in Adults (LADA)
15. (US ONLY) History or current evidence of hematologic condition that would make HbA1c uninterpretable including:

    15.1. Grade 1 anemia, defined as: Hemoglobin (Hb) < Lower Limit of Normal (LLN) - 10.0 g/dL or < LLN - 6.2 mmol/L or < LLN - 100 g/L

    15.2. Hemoglobinopathy, with the exception of sickle cell trait or thalassemia minor; or chronic or recurrent hemolysis

    15.3. Donation of blood or blood products to a blood bank, blood transfusion or participation in a clinical study requiring withdrawal of > 400 mL of blood during the 90 days prior to the Screening visit

    15.4. Significant iron deficiency anemia

    15.5. Heart malformations or Vaso-Occlusive Crisis (VOC) leading to increased turnover of erythrocytes
16. (US ONLY) Current evidence of hypertension defined as the mean (average) of Diastolic Blood Pressure (DBP) > 89 mm Hg or Systolic Blood Pressure (SBP) > 129 mm Hg based on 3 consecutive readings at least 2 minutes apart
17. (US ONLY) History or current evidence of active drug, chemical or alcohol dependency.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Change in stimulated C-peptide response during the first two hours of a mixed meal tolerance test (MMTT) from baseline to 48 weeks between IMCY-0098 and placebo groups | From baseline to 48 weeks
  The area under the stimulated C-peptide response curve over the first two hours of a MMTT

SECONDARY OUTCOMES:
Changes in stimulated C-peptide response during the first two hours of a MMTT for the two doses of IMCY-0098 versus placebo | From baseline to 24 months
  The area under the stimulated C-peptide response curve over the first two hours of a MMTT
Difference in Dried Blood Spots (DBS) fasted C-peptide between treatment and placebo groups | From baseline to 48 weeks
  DBS C-peptide measurements
Changes in DBS C-peptide measurements at each visit comparing each dose with placebo | From baseline to 24 months
  The DBS C-peptide responses at each visit
Effects of each dose of IMCY-0098 on HbA1c | From baseline to 24 months
  Change in HbA1c
Effects of each dose of IMCY-0098 on hypoglycaemic events | From baseline to 24 months
  Number of treatment-emergent severe hypoglycaemic episodes
Effects of each dose of IMCY-0098 on diabetic ketoacidosis (DKA) episodes | From baseline to 24 months
  Number of treatment-emergent episodes of DKA
Effects of each dose of IMCY-0098 on daily total insulin dose | From baseline to 24 months
  Change in insulin requirements as the daily total dose (three days average) in units per kg body weight
Effects of each dose of IMCY-0098 on Continuous Glucose Monitoring (CGM) measures | From baseline to 24 months
  CGM time in range (70-180 mg/dL, 3.9- 10.0 mmol/L), time above range (>180 mg/dL, >10.0 mmol/L), time below range (<70 mg/dL, < 3.9 mmol/L) during 10 days compared to the reference period (first 10 days after randomization)
Impact of IMCY-0098 at each dose on autoantibodies against GAD65, IA 2, ZnT8 and insulin over time | From baseline to 24 months
  Change in T1D associated autoantibodies (GADA, IAA, IA-2A and ZnT8A)
To evaluate the safety features of IMCY-0098 during treatment period | Up to 7 days after the last dose
  Occurrence, intensity and relationship of any listed injection site and systemic AEs during a 7-day follow-up period after each dose
To evaluate the safety features of IMCY-0098 during the whole study duration | Up to 48 weeks
  Occurrence, intensity and relationship of any unlisted injection site and AEs and occurrence and relationship of all SAEs and abnormality in physical examination, vital signs, 12-lead ECG
To evaluate the safety features of IMCY-0098 on lymphocytes ratio | Up to 48 weeks
  Measure of CD4+/CD8+ lymphocytes ratio

CONTACTS AND LOCATIONS:
Overall Officials: Jean Van Rampelbergh, Study Director — Imcyse SA
Locations (29):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Barbara Davis Center, Aurora, Colorado
  - University of Chicago, Chicago, Illinois
  - Joslin Diabetes Center, Boston, Massachusetts
- Australia (4):
  - Princess Alexandra Hospital, Brisbane
  - Royal Melbourne Hospital, Melbourne
  - St. Vincent's Hospital, Melbourne
  - Royal North Shore Hospital, Sydney
- Belgium (3):
  - Université Libre de Bruxelles - Hôpital Erasme - ULB, Brussels
  - UZ Brussels, Brussels
  - Katholieke Universiteit Leuven UZ Gasthuisberg, Leuven
- Italy (2):
  - Ospedale San Raffaele S.r.l., Milan
  - AOU Pisana - Ospedale Cisanello, Pisa
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kauno Klinikos, Kaunas
  - Klaipeda university hospital, Klaipėda
  - Vilnius university hospital Santaros klinikos, Vilnius
- UMC - University Children's Hospital, Ljubljana, Slovenia
- Department of clinical sciences, CRC/Malmö, Lund University, Lund, Sweden
- United Kingdom (11):
  - Addenbrooke's Hospital, Cambridge
  - University Hospital of Wales, Cardiff
  - Royal Infirmary of Edinburgh, Edinburgh
  - Royal Devon and Exeter Hospital, Exeter
  - St James´s University Hospital, Leeds
  - Leicester General Hospital, Leicester
  - Guy's and St Thomas' Hospital, London
  - Royal London Hospital, London
  - St George's Hospital, London
  - Royal Victoria Infirmary, Newcastle
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No